CLINICAL TRIAL: NCT07165353
Title: Virtual Walking With Habitual Feedback to Reduce Chronic Neuropathic Pain in Individuals With Spinal Cord Injury
Brief Title: Virtual Walking to Reduce Chronic Neuropathic Pain in Subjects With SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-17
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries (SCI); Neuropathic Pain Due to Spinal Cord Injury
Keywords: neuropathic pain; virtual walking; virtual reality; spinal cord injury pain; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants will receive virtual walking (VW) therapy with a personalized avatar. Using a green screen setup, a live video of the participant's upper body is combined with pre-recorded walking legs to create a full-body walking illusion, displayed on a large projection screen in a forest environment. The participant will be seated in a modified wheelchair that tilts 2° to each side to simulate pelvic movement during walking.
  Interventions: Behavioral: Virtual Walking
- Group 2 (Sham Comparator): Participants will receive virtual walking (VW) therapy without an avatar. The screen will display only a moving forest environment, and the wheelchair tilt will be omitted. This condition serves as a sham intervention, matching Group 1 in session number, duration, and procedure, but without the visual and vestibular walking components.
  Interventions: Behavioral: Sham Virtual Walking
- Control Group (No Intervention): Participants will receive standard medical pain management only. They will not take part in virtual walking therapy but will complete the pain diary and questionnaires at the scheduled assessment time points.

INTERVENTIONS:
Behavioral: Virtual Walking — This virtual walking therapy uses a life-sized video avatar of the participant walking through a forest environment. A green screen setup combines a live video of the participant's upper body with pre-recorded walking legs, creating a full-body walking illusion. The participant is seated in a modified wheelchair that tilts 2° to each side to mimic pelvic movement during walking. This approach differs from the sham condition (Group 2), which displays only the moving forest without an avatar or wheelchair tilt, and from the standard care group (Group 3), which receives no virtual walking therapy.
  Arms: Group 1
Behavioral: Sham Virtual Walking — Participants view a moving forest environment on a large projection screen for 10 sessions over 2 weeks (each up to 20 minutes). No avatar of the participant is displayed, and the wheelchair tilt function is disabled. This differs from the experimental intervention (Group 1), which includes a life-sized walking avatar and wheelchair tilt to mimic pelvic movement, and from the standard care group (Group 3), which receives no virtual walking therapy.
  Arms: Group 2

SUMMARY:
About 70% of people with a spinal cord injury in Switzerland have chronic pain that lasts more than 3 to 6 months. This pain can be caused by muscle or joint problems, or by nerve damage (neuropathic pain). Neuropathic pain is often hard to treat, and current treatments may cause side effects or not work well.

This study will test whether virtual walking from different visual perspectives can reduce chronic neuropathic pain and improve quality of life after spinal cord injury. We will also compare which perspective works best.

To better understand how the training works, we will use two tests-quantitative sensory testing (QST) and contact heat-evoked potentials (CHEPs)-to measure changes in the pain and nerve systems.

DETAILED DESCRIPTION:
Chronic pain conditions are highly prevalent in the Swiss spinal cord injury (SCI) population with a prevalence of 73% (Müller et al., 2017). Most of those individuals show multiple pain modalities (neuropathic, nociceptive and unknown pain type) (Mahnig et al., 2016; Siddall et al., 2003). For example, Mahnig et al. (2016) reported prevalences of 79% neuropathic and 61% nociceptive pain in individuals with SCI seen in a pain clinic. The current practice of pharmacological first- and second-line treatments comes along with many side effects and unsatisfactory results (Finnerup et al., 2015). This is because the underlying biology of chronic neuropathic pain (NeP) and the mechanisms that lead to chronification of pain are highly complex and not fully understood. Latest research suggests that chronification of pain is associated with anatomical and functional reorganization of the brain (Reckziegel et al., 2019; Wrigley et al., 2009). More specifically, cortical grey matter density changes and neuroanatomical reorganization of the primary somatosensory cortex are discussed as factors associated with pain chronification. Additional mechanisms proposed to explain NeP after SCI include spinal cord plasticity, supraspinal reorganization, and increased neuronal excitability of dorsal horn neurons (Finnerup, 2013).

MRI data show, that there is a correlation between the grade of cortical reorganisation and pain intensity in people with complete SCI (Gustin et al., 2023). However, it is unclear whether there is a systematic influence of the severity of the SCI lesion, graded by the American Spinal Injury Association (ASIA) Impairment Scale (complete or incomplete SCI), on pain intensity.

Alongside with studies about pain mechanisms and improved pharmaceutical treatment, non-invasive and non-pharmacological alternative treatments with minimal side effects have been investigated, such as, for example virtual reality (VR). Changes of pain perception due to VR interventions in individuals with neuropathic spinal cord injury pain (SCIP) are described in the literature (Eick & Richardson, 2015; Kumru et al., 2013; Moseley, 2007; Özkul et al., 2015; Soler et al., 2010; Trost et al., 2022). Recent reviews have shown good short-term effects of VR in the treatment of SCIP (Chi et al., 2019; de Araújo et al., 2019). However, there is lack of evidence from randomized controlled trials.

Chronic pain in SCI is often modulated by psycho-social factors such as depression, anxiety, extent of social support and pain catastrophising (Braunwalder et al., 2022; Braunwalder et al., 2021; Müller et al., 2017; Wollaars et al., 2007). Data about the influence of psycho-social factors on VR therapy are only reported for VR therapy in first person perspective (Trost et al., 2022). Data about the influence of psycho-social factors third person perspective are not available.

Recently, a virtual walking (VW) treatment protocol in third person perspective inclusive an additional haptic feedback modality (controlled movement of the wheelchair seat to improve the walking immersion) has been set up and evaluated within a feasibility study with individuals with SCIP, reporting a high level of satisfaction and acceptance of the VW procedure at the Centre for Pain Medicine, Swiss Paraplegic Centre (SPC), Nottwil. In this uncontrolled explorative trial, there was a tendency towards reduced pain intensity and spread of reported pain after VW (Aerni, 2020).

To better understand individual responses to VR and explore underlying pain mechanisms, neurophysiological assessments such as quantitative sensory testing (QST) and contact heat-evoked potentials (CHEPs) are used as biomarkers to identify sensory phenotypes.

To address the challenges of assessing and treating pain following SCI, the systematic evaluation of all somatosensory submodalities is strongly recommended for both pathophysiological research and treatment trials in individuals with SCI-related pain (Finnerup, 2013).

Landmann et al. (2024) demonstrated that QST can identify distinct sensory phenotypes in individuals with neuropathic spinal cord injury pain (SCIP). Furthermore, the combination of QST and CHEPs enables objective and standardized measurement of sensory system alterations, thereby contributing to a better understanding of underlying mechanisms (Opsommer et al., 2021).

The aim of the present study is to evaluate (1) the efficiency of the standardised VW-setting with regard to pain reduction in subjects with complete and incomplete SCI, (2) bio-psycho-social prognostic factors which may influence the efficacy of VR, and (3) the influence of VR on psycho-social characteristics of subjects with SCI and (4) to identify pain and sensory phenotypes in individuals with SCIP and examine whether these phenotypes are associated with differential effects of VR on pain reduction..

ELIGIBILITY:
Inclusion Criteria:

* Sufficient knowledge of German language to understand the instructions, assessments and to fill in questionnaires.
* Age ≥ 18y, ≤ 75y
* Chronic traumatic or non-traumatic SCI (>6 month after SCI) with an SCI severity grade AIS A, B, C or D
* At or below level spinal cord injury neuropathic pain on trunk or lower extremities diagnosed by a neurologist following the ISCIP classification (Bryce et al., 2012) of at least 4/10 intensity on a NRS (Langford et al., 2023)
* Ability to draw with a pen

Exclusion Criteria:

* - Serious psychiatric disorders, which are accompanied by imminent or current acute harm to oneself or others, or which require inpatient psychiatric treatment for other reasons, or other indications of a foreseeable, seriously harmful effect of participation in the study based on the clinical impression from the psychological screening interview
* Participants with a walking ability more than 5 minutes without walking aids
* Pregnancy (anamnestic) in women of child-bearing age (18-49 years)
* Known epilepsy
* neurological disorders (multiple sclerosis, ALS, Guillan-Barré Syndrome, congenital disorders, polyneuropathy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a clinically meaningful reduction in average pain intensity | 15 weeks
  The primary outcome is the percentage of participants achieving a reduction of ≥1 point on the Numeric Rating Scale (NRS; 0 = no pain, 10 = worst imaginable pain) for average pain intensity. Pain intensity is assessed daily using a pain diary over one week, measured at 4 weeks and 12 weeks after the end of treatment, compared to baseline (1 week before treatment start).

SECONDARY OUTCOMES:
Change in pain distribution | Baseline (1 week before intervention) to 2, 3, 4, 7, and 15 weeks after start of intervention
  Extent of pain area (size in pixels and percentage of total body chart) indicated by the participant on a standardized pain drawing.
Change in pain distribution | Baseline (1 week before intervention) to 2, 3, 4, 7, and 15 weeks after start of intervention
  Average pain intensity measured daily using a pain diary and the Numeric Rating Scale (NRS; 0 = no pain, 10 = worst imaginable pain) over one week at each time point, compared to baseline.
Pain interference, diagnosis, type, and duration | Baseline, 4 and 12 weeks post-treatment
  Measured using the Spinal Cord Injury Pain Basic Data Set (SCIP-BDS 3.0).
Neuropathic pain quality | Baseline, 4 and 12 weeks post-treatment
  Measured using the Neuropathic Pain Symptom Inventory (NPSI).
Severity of chronic pain | Baseline, 4 and 12 weeks post-treatment
  Measured using the Chronic Pain Grading Scale (CPGS).
Pain chronicity | Baseline, 4 and 12 weeks post-treatment
  Measured using the Mainz Pain Staging System (MPSS).
General health-related quality of life | Baseline, 4 and 12 weeks post-treatment
  Measured using the Veterans RAND 12 Item Health Survey (VR-12).
General well-being | Baseline, 4 and 12 weeks post-treatment
  Measured using the Spinal Cord Injury Quality of Life Basic Data Set (SCI-QoL-BDS) and the Marburg Questionnaire on Habitual Well-being (FW-7).
Pain catastrophizing | Baseline, 4 and 12 weeks post-treatment
  Measured using the Pain Catastrophizing Scale (PCS).
Depression, anxiety, and stress | Baseline, 4 and 12 weeks post-treatment
  Measured using the Depression Anxiety and Stress Scale (DASS).
Subjective impression of change | 4 and 12 weeks post-treatment
  Measured using the Patient Global Impression of Change (PGIC).
Experienced emotions | Baseline, 4 and 12 weeks post-treatment
  Measured using the Scales for the Assessment of Emotional Experience (SEE).
Positive outcomes after traumatic events | Baseline, 4 and 12 weeks post-treatment
  Measured using the Posttraumatic Growth Inventory (PTGI).
Posttraumatic stress disorder | Baseline, 4 and 12 weeks post-treatment
  Measured using the International Trauma Questionnaire (ITQ).
Clinical data | Baseline
  Includes age, gender, age at injury, lesion level, completeness of lesion, grade of motor function, concomitant injuries, pain quality, and medication, obtained from clinical records or assessed by the International SCI Core Data Set (I-SCI-CDS)
Severity grades of SCI | Baseline
  Assessed using the American Spinal Injury Association (ASIA) Impairment Scale (AIS A-D)

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Landmann, KD Dr. med., Principal Investigator — Schweizer Paraplegiker Zentrum Nottwil
Locations (1):
- Schweizer Paraplegiker Zentrum Nottwil, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the informed consent and ethics approval do not include permission for data sharing, and to ensure protection of participant privacy.

REFERENCES:
- [Background] Mahnig S, Landmann G, Stockinger L, Opsommer E. Pain assessment according to the International Spinal Cord Injury Pain classification in patients with spinal cord injury referred to a multidisciplinary pain center. Spinal Cord. 2016 Oct;54(10):809-815. doi: 10.1038/sc.2015.219. Epub 2016 Jan 12. PMID 26754471
- [Background] Finnerup NB, Attal N, Haroutounian S, McNicol E, Baron R, Dworkin RH, Gilron I, Haanpaa M, Hansson P, Jensen TS, Kamerman PR, Lund K, Moore A, Raja SN, Rice AS, Rowbotham M, Sena E, Siddall P, Smith BH, Wallace M. Pharmacotherapy for neuropathic pain in adults: a systematic review and meta-analysis. Lancet Neurol. 2015 Feb;14(2):162-73. doi: 10.1016/S1474-4422(14)70251-0. Epub 2015 Jan 7. PMID 25575710
- [Background] Finnerup NB. Pain in patients with spinal cord injury. Pain. 2013 Dec;154 Suppl 1:S71-S76. doi: 10.1016/j.pain.2012.12.007. Epub 2012 Dec 22. PMID 23375163
- [Result] Wydenkeller S, Maurizio S, Dietz V, Halder P. Neuropathic pain in spinal cord injury: significance of clinical and electrophysiological measures. Eur J Neurosci. 2009 Jul;30(1):91-9. doi: 10.1111/j.1460-9568.2009.06801.x. Epub 2009 Jun 25. PMID 19558605
- [Result] Wrigley PJ, Press SR, Gustin SM, Macefield VG, Gandevia SC, Cousins MJ, Middleton JW, Henderson LA, Siddall PJ. Neuropathic pain and primary somatosensory cortex reorganization following spinal cord injury. Pain. 2009 Jan;141(1-2):52-9. doi: 10.1016/j.pain.2008.10.007. Epub 2008 Nov 21. PMID 19027233
- [Result] Widerstrom-Noga E, Biering-Sorensen F, Bryce TN, Cardenas DD, Finnerup NB, Jensen MP, Richards JS, Rosner J, Taylor J. The international spinal cord injury pain basic data set (version 3.0). Spinal Cord. 2023 Oct;61(10):536-540. doi: 10.1038/s41393-023-00919-w. Epub 2023 Jul 25. PMID 37491608
- [Result] Von Korff M, Ormel J, Keefe FJ, Dworkin SF. Grading the severity of chronic pain. Pain. 1992 Aug;50(2):133-149. doi: 10.1016/0304-3959(92)90154-4. PMID 1408309
- [Result] Turk DC, Dworkin RH, Allen RR, Bellamy N, Brandenburg N, Carr DB, Cleeland C, Dionne R, Farrar JT, Galer BS, Hewitt DJ, Jadad AR, Katz NP, Kramer LD, Manning DC, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robinson JP, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Witter J. Core outcome domains for chronic pain clinical trials: IMMPACT recommendations. Pain. 2003 Dec;106(3):337-345. doi: 10.1016/j.pain.2003.08.001. PMID 14659516
- [Result] Trost Z, Anam M, Seward J, Shum C, Rumble D, Sturgeon J, Mark V, Chen Y, Mitchell L, Cowan R, Perera R, Richardson E, Richards S, Gustin S. Immersive interactive virtual walking reduces neuropathic pain in spinal cord injury: findings from a preliminary investigation of feasibility and clinical efficacy. Pain. 2022 Feb 1;163(2):350-361. doi: 10.1097/j.pain.0000000000002348. PMID 34407034
- [Result] Sommer C, Richter H, Rogausch JP, Frettloh J, Lungenhausen M, Maier C. A modified score to identify and discriminate neuropathic pain: a study on the German version of the Neuropathic Pain Symptom Inventory (NPSI). BMC Neurol. 2011 Aug 23;11:104. doi: 10.1186/1471-2377-11-104. PMID 21861889
- [Result] Richardson EJ, McKinley EC, Rahman AKMF, Klebine P, Redden DT, Richards JS. Effects of virtual walking on spinal cord injury-related neuropathic pain: A randomized, controlled trial. Rehabil Psychol. 2019 Feb;64(1):13-24. doi: 10.1037/rep0000246. Epub 2018 Nov 8. PMID 30407030
- [Result] Pfau DB, Krumova EK, Treede RD, Baron R, Toelle T, Birklein F, Eich W, Geber C, Gerhardt A, Weiss T, Magerl W, Maier C. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): reference data for the trunk and application in patients with chronic postherpetic neuralgia. Pain. 2014 May;155(5):1002-1015. doi: 10.1016/j.pain.2014.02.004. Epub 2014 Feb 10. PMID 24525274
- [Result] Ozkul C, Kilinc M, Yildirim SA, Topcuoglu EY, Akyuz M. Effects of visual illusion and transcutaneous electrical nerve stimulation on neuropathic pain in patients with spinal cord injury: A randomised controlled cross-over trial. J Back Musculoskelet Rehabil. 2015;28(4):709-19. doi: 10.3233/BMR-140573. PMID 25502348
- [Result] Opsommer E, Korogod N, Stockinger L, Landmann G. Multimodal sensory evaluation of neuropathic spinal cord injury pain: an experimental study. Spinal Cord. 2021 Aug;59(8):842-854. doi: 10.1038/s41393-020-00607-z. Epub 2021 Jan 14. PMID 33446934
- [Result] Moseley LG. Using visual illusion to reduce at-level neuropathic pain in paraplegia. Pain. 2007 Aug;130(3):294-298. doi: 10.1016/j.pain.2007.01.007. Epub 2007 Mar 1. PMID 17335974
- [Result] Magerl W, Krumova EK, Baron R, Tolle T, Treede RD, Maier C. Reference data for quantitative sensory testing (QST): refined stratification for age and a novel method for statistical comparison of group data. Pain. 2010 Dec;151(3):598-605. doi: 10.1016/j.pain.2010.07.026. Epub 2010 Oct 20. PMID 20965658
- [Result] Maercker, A. L., R. (2001). Persönliche Reifung (Personal Growth) durch Belastungen und Traumata. Diagnostica, VOL.47,NO.3. https://doi.org/https://doi.org/10.1026//0012-1924.47.3.153
- [Result] Langford DJ, Baron R, Edwards RR, Gewandter JS, Gilron I, Griffin R, Kamerman PR, Katz NP, McDermott MP, Rice ASC, Turk DC, Vollert J, Dworkin RH. What should be the entry pain intensity criteria for chronic pain clinical trials? An IMMPACT update. Pain. 2023 Sep 1;164(9):1927-1930. doi: 10.1097/j.pain.0000000000002930. Epub 2023 Jun 7. No abstract available. PMID 37288944
- [Result] Kumru H, Soler D, Vidal J, Navarro X, Tormos JM, Pascual-Leone A, Valls-Sole J. The effects of transcranial direct current stimulation with visual illusion in neuropathic pain due to spinal cord injury: an evoked potentials and quantitative thermal testing study. Eur J Pain. 2013 Jan;17(1):55-66. doi: 10.1002/j.1532-2149.2012.00167.x. Epub 2012 May 18. PMID 22610590
- [Result] Kirshblum SC, Burns SP, Biering-Sorensen F, Donovan W, Graves DE, Jha A, Johansen M, Jones L, Krassioukov A, Mulcahey MJ, Schmidt-Read M, Waring W. International standards for neurological classification of spinal cord injury (revised 2011). J Spinal Cord Med. 2011 Nov;34(6):535-46. doi: 10.1179/204577211X13207446293695. No abstract available. PMID 22330108
- [Result] Kazis LE, Miller DR, Skinner KM, Lee A, Ren XS, Clark JA, Rogers WH, Spiro A 3rd, Selim A, Linzer M, Payne SM, Mansell D, Fincke RG. Patient-reported measures of health: The Veterans Health Study. J Ambul Care Manage. 2004 Jan-Mar;27(1):70-83. doi: 10.1097/00004479-200401000-00012. PMID 14717468
- [Result] Gustin SM, Bolding M, Willoughby W, Anam M, Shum C, Rumble D, Mark VW, Mitchell L, Cowan RE, Richardson E, Richards S, Trost Z. Cortical Mechanisms Underlying Immersive Interactive Virtual Walking Treatment for Amelioration of Neuropathic Pain after Spinal Cord Injury: Findings from a Preliminary Investigation of Thalamic Inhibitory Function. J Clin Med. 2023 Sep 4;12(17):5743. doi: 10.3390/jcm12175743. PMID 37685810
- [Result] de Araujo AVL, Neiva JFO, Monteiro CBM, Magalhaes FH. Efficacy of Virtual Reality Rehabilitation after Spinal Cord Injury: A Systematic Review. Biomed Res Int. 2019 Nov 13;2019:7106951. doi: 10.1155/2019/7106951. eCollection 2019. PMID 31828120
- [Result] Christen D, Killikelly C, Maercker A, Augsburger M. Item Response Model Validation of the German ICD-11 International Trauma Questionnaire for PTSD and CPTSD. Clin Psychol Eur. 2021 Dec 23;3(4):e5501. doi: 10.32872/cpe.5501. eCollection 2021 Dec. PMID 36398291
- [Result] Charlifue S, Post MW, Biering-Sorensen F, Catz A, Dijkers M, Geyh S, Horsewell J, Noonan V, Noreau L, Tate D, Sinnott KA. International Spinal Cord Injury Quality of Life Basic Data Set. Spinal Cord. 2012 Sep;50(9):672-5. doi: 10.1038/sc.2012.27. Epub 2012 Mar 27. PMID 22450884
- [Result] Braunwalder C, Muller R, Kunz S, Tough H, Landmann G, Fekete C. Psychosocial resources and chronic pain in individuals with spinal cord injury: evidence from the second Swiss national community survey. Spinal Cord. 2021 Apr;59(4):410-418. doi: 10.1038/s41393-020-00577-2. Epub 2020 Nov 19. PMID 33214625
- [Result] Braunwalder C, Ehrmann C, Hodel J, Muller R, von Matt D, Fekete C. Pain Trajectories During Initial Rehabilitation After Spinal Cord Injury: Do Psychosocial Resources and Mental Health Predict Trajectories? Arch Phys Med Rehabil. 2022 Jul;103(7):1294-1302. doi: 10.1016/j.apmr.2022.01.149. Epub 2022 Feb 11. PMID 35157891
- [Result] Bouhassira D, Branders S, Attal N, Fernandes AM, Demolle D, Barbour J, Ciampi de Andrade D, Pereira A. Stratification of patients based on the Neuropathic Pain Symptom Inventory: development and validation of a new algorithm. Pain. 2021 Apr 1;162(4):1038-1046. doi: 10.1097/j.pain.0000000000002130. PMID 33136982
- [Result] Biering-Sorensen F, Charlifue S, Chen Y, New PW, Noonan V, Post MWM, Rupp R, Vogel L. International Spinal Cord Injury Core Data Set (version 3.0)-including standardization of reporting. Spinal Cord. 2023 Jan;61(1):65-68. doi: 10.1038/s41393-022-00862-2. Epub 2022 Oct 28. PMID 36307730
- [Result] Schmerz.) Behr, M. B., M. . (2004). Skalen zum Erleben von Emotionen (SEE). Göttingen: Hogrefe.
- [Result] Aerni, M. (2020). Machbarkeitsstudie: Virtual walking bei Personen mit neuropathischen Schmerzen infolge Querschnittlähmung. . Master thesis, University of applied sciences Zurich.